CLINICAL TRIAL: NCT03257098
Title: An Interventional, Single Arm, Multicenter, Phase I/IIa Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-CVU on Wound Healing of Chronic Venous Ulcer (CVU)
Brief Title: Allogeneic ABCB5-positive Stem Cells for Treatment of CVU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Ticeba GmbH (Industry); Granzer Regulatory Consulting & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: allo-APZ2-CVU-II-01
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Skin Ulcer Venous Stasis Chronic
Keywords: Chronic Venous Ulcer; ABCB5; Allogeneic; Mesenchymal stem cells; varicose ulcer; skin ulcer; advanced therapy medicinal product; somatic cell therapy; phase I/IIa
MeSH Terms: conditions — Varicose Ulcer; Skin Ulcer

STUDY DESIGN:
Intervention Model Description: Interventional, single arm, multicenter, phase I/IIa clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allo-APZ2-CVU (Experimental): Application of IMP on patients wound
  Interventions: Biological: allo-APZ2-CVU

INTERVENTIONS:
Biological: allo-APZ2-CVU — Suspension of ABCB5-positive mesenchymal stem cells

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring the wound size reduction of Chronic Venous Ulcers) and safety (by monitoring adverse events) of the medicinal product to be studied after two applications on the wound surface in patients with Chronic Venous Ulcers.

DETAILED DESCRIPTION:
This is an interventional, single arm, phase I/IIa clinical trial to investigate the efficacy and safety of allogeneic ABCB5-positive mesenchymal stem cells (MSCs) on wound healing in patients with chronic venous ulcer (CVU). Allogeneic MSCs will be isolated ex vivo and will be expanded in vitro. The IMP incorporating the ABCB5-positive MSCs will then be applied on the wound surface of CVU under local anesthesia (on Day 0 and Week 6.1).

Wound measurements from Visit (V) 2 and V9 will be used to determine the cell amount for the IMP treatments on V3 and V10, respectively.

Patients are followed up for efficacy for 3 months which allows to distinguish actual wound healing from transient wound coverage.

The wound healing process will be documented by standardized photography. The wound size evaluation will start on the day of the first change of wound dressing. The quality of the wound healing process will be assessed on the basis of formation of granulation tissue, epithelialization and wound exudation.

Pain will be assessed using a numerical rating scale and quality of life will be investigated with standardized and validated questionnaires. To assess long-term safety of allo-APZ2-CVU three follow-up visits at Months 6, 9 and 12 after the first IMP applications are included.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 35 to 85 years;
2. Chronic venous leg ulcer (as defined by the current AWMF guidelines: therapy resistant ulcer that shows no improvement within 3 months despite of optimal phlebological therapies or is not healed within 12 months) diagnosed by doppler ultrasonography (DUS), ankle brachial index (ABI, 0.9-1.3), physical examination and dermatological review;
3. Wound size of target ulcer between 1.5 and 100 cm2 measured by a standardized photography at the screening visits (Visit 1 and Visit 2);
4. Wound location below knee;
5. If patients are suffering from 2 or more ulcers at the same extremity, the target ulcer has to be separated by a minimum bridge of 1 cm of epithelialized skin from other ulcers (the largest ulcer should be the target ulcer, if not decided otherwise at discretion of the investigator; the target ulcer is defined at Visit 1);
6. Body mass index (BMI) between 20 and 45 kg/m²;
7. Patients understand the nature of the procedure and are providing written informed consent prior to any clinical trial procedure;
8. Women of childbearing potential must have a negative blood pregnancy test at Visit 1
9. Women of childbearing potential and their partner must be willing to use highly effective contraceptive methods during the course of the clinical trial.

Exclusion Criteria:

1. Evidence of the ulcer extending to the underlying muscle, tendon, or bone;
2. Current use of systemic steroid medication above Cushing threshold dose (>7.5 mg/d prednisone or equivalent);
3. Diabetes mellitus that has to be evaluated by blood test (Haemoglobin A1c [HbA1c] >7.5%);
4. Peripheral Artery Disease (PAD) including claudication with need of treatment;
5. Acute deep vein thrombosis (maximum 30 days from diagnosis) or a still untreated deep vein thrombosis;
6. Unable to tolerate leg ulcer compression bandage;
7. Infection of the target ulcer requiring treatment as judged clinically;
8. Any chronic dermatological disorders diagnosed at the investigator's discretion;
9. Skin disorders, unrelated to the ulcer, that are present adjacent to the target wound;
10. Current use of medications that influence wound healing: systemic immunosuppressives, cytotoxic medicinal products, and systemic steroids (above Cushing-threshold level);
11. Known abuse of alcohol, drugs, or medicinal products;
12. Cancerous or pre-cancerous lesions adjacent to the target wound;
13. Patients anticipated to be unwilling or unable to comply with the requirements of the protocol;
14. Pregnant or lactating women;
15. Systemic infectious disease diagnosed by serology testing human immunodeficiency virus (HIV˗1, HIV-2);
16. Any known allergies to components of the IMP;
17. Prior surgical procedures such as bypass or mesh-graft treatment within 2 months prior to Visit 1;
18. Patients with significant ulcer healing or wound size enlargement of more than 25% at Visit 2 compared to Visit 1;
19. Treatment of target ulcer with active wound care agents (e.g. iruxol, local antibiotics or silver dressings), which have not been paused 14 days before IMP application;
20. Current or previous (within 30 days of enrollment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
21. Previous participation in this clinical trial (except for screening failures due to an inclusion or exclusion criterion);
22. Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
23. Employees of the sponsor, or employees or relatives of the investigator.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Percentage of wound size reduction | Week 12 post baseline, or last available post-baseline measurement if the Week 12 measurement is missing
  Percentage of wound size reduction at Week 12, or last available post-baseline measurement of Weeks 6, 8 or 10 if the Week 12 measurement is missing (last observation carried forward [LOCF]).
Assessment of adverse event (AE) occurrence | Up to 12 months
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Percentage of wound size reduction | Weeks 2, 3, 4, 6, 6.1, 6.2, 8, 10, and 12 (without LOCF);
Absolute wound size reduction | Weeks 2, 3, 4, 6, 6.1, 6.2, 8, 10, and 12
Proportion of patients achieving complete wound closure | Weeks 2, 3, 4, 6, 8, 10, 12, and at any time point
Time to first complete wound closure | A priori specification not possible; between baseline and week 12 post baseline
Proportion of patients achieving 30% wound closure | Weeks 2, 3, 4, 6, 6.1, 6.2, 8, 10, 12, and at any time point
Time to first 30% wound closure | A priori specification not possible; between baseline and week 12 post baseline
Epithelialization | Weeks 2, 3, 4, 6, 6.1, 6.2, 8, 10, and 12
Assessment of further wound healing parameters: formation of granulation tissue and wound exudation | Visit 3 and Visit 10 before IMP application, Days 1 to 3 and 8, Weeks 2, 3, 4, 6, 6.2, 8, 10, and 12
Pain assessment as per numerical rating scale (NRS) | Days 0, 1 to 3 and 8, Weeks 2, 3, 4, 6, 6.1, 6.2, 8, 10, and 12
Assessment of quality of life (QoL) using the short form 36 (SF-36) questionnaire | Day 0 and Weeks 4, 8 and 12
Assessment of dermatology-specific quality of life based on the Dermatology Life Quality Index (DLQI) questionnaire | Day 0 and Weeks 4, 8 and 12
Physical examination and vital signs at Week 6.1 and Week 12 | Week 6.1 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kerstan, Dr., Principal Investigator — Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Würzburg
Locations (9):
- Germany (9):
  - Venenzentrum der Dermatologischen und Gefäßchirurgischen Kliniken, Kliniken der Ruhr-Universität Bochum im St. Maria Hilf Krankenhaus, Bochum
  - Universitätsklinikum Erlangen, Hautklinik, Erlangen
  - Klinik und Poliklinik für Hautkrankheiten, Universitätsmedizin Greifswald, Greifswald
  - Klinische Forschung Hamburg GmbH, Dermatologie / Allergologie, Hamburg
  - pro scientia med im Mare Klinikum; Department Klinische Forschung und Entwicklung, Kiel
  - Universitätsklinikum Münster, Klinik für Hautkrankheiten, Allgemeine Dermatologie und Venerologie, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Universitätsklinikum Ulm, Klinik für Dermatologie und Allergologie, Ulm
  - Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerstan A, Niebergall-Roth E, Esterlechner J, Schroder HM, Gasser M, Waaga-Gasser AM, Goebeler M, Rak K, Schrufer P, Endres S, Hagenbusch P, Kraft K, Dieter K, Ballikaya S, Stemler N, Sadeghi S, Tappenbeck N, Murphy GF, Orgill DP, Frank NY, Ganss C, Scharffetter-Kochanek K, Frank MH, Kluth MA. Ex vivo-expanded highly pure ABCB5+ mesenchymal stromal cells as Good Manufacturing Practice-compliant autologous advanced therapy medicinal product for clinical use: process validation and first in-human data. Cytotherapy. 2021 Feb;23(2):165-175. doi: 10.1016/j.jcyt.2020.08.012. Epub 2020 Oct 1. PMID 33011075